CLINICAL TRIAL: NCT00161473
Title: Alzheimer's in Long-Term Care--Treatment for Agitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16508-A; 5R01AG018644 (NIH); 5P50AG005136 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-06

CONDITIONS: Alzheimer Disease; Psychomotor Agitation
Keywords: double-blind; treatment; prazosin
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prazosin (Active Comparator)
  Interventions: Drug: prazosin
- placebo (inert substance) (Placebo Comparator)
  Interventions: Drug: placebo (inert substance)

INTERVENTIONS:
Drug: prazosin — Participants taking prazosin. Prazosin was administered as 1 or 2 mg capsules. Doses were initiated at 1 mg at bedtime. Titration based on tolerability was conducted up to a dose of 2 mg in the morning plus 4mg at bedtime.
  Duration was 8 weeks.
  Other Names: Minipress
  Arms: prazosin
Drug: placebo (inert substance) — Placebo is an inert substance used as a standard comparator in clinical pharmacologic trials. Duration is 8 weeks.
  Arms: placebo (inert substance)

SUMMARY:
The purpose of this study is to see if a medication called prazosin is useful in the treatment of agitation and aggression in persons with Alzheimer's disease (AD) and other types of dementia in late life.

DETAILED DESCRIPTION:
Although the occurrence of disruptive agitation behaviors likely are influenced by environmental/ interpersonal factors, it is also likely that behaviorally relevant neurobiologic abnormalities lower the threshold for the expression of such behavior in Alzheimer's disease. Because of the success prazosin has had in the treatment of Posttraumatic Stress Disorder, it is thought that it could be used similarly with disruptive agitation. Originally designed to evaluate Alzheimer's disease patients in nursing homes, the study now includes outpatients. It is a 9-week placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* No age limit
* probable/possible Alzheimer's disease diagnosis
* disruptive agitated behaviors (e.g., irritability, aggression, uncooperativeness, pacing)
* no hypotension
* no concurrent use of alpha-1-blockers
* no delirium, schizophrenia, mania, psychotic symptoms.

Exclusion Criteria:

* Cardiovascular: unstable angina, recent myocardial infarction, second or third degree atrioventricular (AV) block, preexisting hypotension (systolic blood pressure less than 110) or orthostatic hypotension
* Other medical exclusions: chronic renal or hepatic failure, or any unstable medical condition
* Exclusionary medications: current treatment with prazosin, other alpha-1-blockers
* Current enrollment in a separate investigational drug trial
* Psychoactive medications: subjects may be psychoactive medication-free or be partial responders (by subjective assessment of referring health care professional) to one psychoactive medication from any of the following classes: antipsychotics, anticonvulsants, mood stabilizers, antidepressants, benzodiazepines, or buspirone. Partial response is defined as some improvement in agitated behavior but persistence of agitated behaviors severe enough to cause patient distress and/or difficulty with caregiving. Although not formally rated, this improvement is equivalent to a Clinical Global Impression of Change (CGIC) rating of no more than minimal improvement (improvement is noticed by not enough to improve patient function or caregiver's practical management of the patient).
* Psychiatric/behavioral: lifetime schizophrenia; current delirium, mania, depression, or uncontrolled persistent distressing psychotic symptoms (hallucinations, delusions), substance abuse, panic disorder, or any behavior which poses an immediate danger to patient or others or which results in the patient being too uncooperative to meet the requirements of study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine R Peskind, MD, Principal Investigator — Veterans Affairs Puget Sound Health Care System
Locations (1):
- Veterans Affairs Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Result] Wang LY, Shofer JB, Rohde K, Hart KL, Hoff DJ, McFall YH, Raskind MA, Peskind ER. Prazosin for the treatment of behavioral symptoms in patients with Alzheimer disease with agitation and aggression. Am J Geriatr Psychiatry. 2009 Sep;17(9):744-51. doi: 10.1097/JGP.0b013e3181ab8c61. PMID 19700947

RESULTS

PARTICIPANT FLOW:
Groups:
- Prazosin: Participants taking prazosin. Prazosin was administered as 1 or 2 mg capsules. Doses were initiated at 1 mg at bedtime. Titration based on tolerability was conducted up to a dose of 2 mg in the morning plus 4mg at bedtime.
- Placebo: Placebo is an inert substance used as a standard comparator in clinical pharmacologic trials.
Period: Overall Study
Arm/Group | Prazosin | Placebo
Started | 12 | 12
Completed | 7 | 6
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 12 | 12 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 83.2 (11.5) | 78.1 (10.8) | 80.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Clinical Global Impression of Change (CGIC) at Last Observation
Description: The Clinical Global Impression of Change (CGIC) is a 7 point scale, where 1 indicates "markedly improved," 4 indicates "no change," and 7 indicates "markedly worse."
Time Frame: Week 8
Population: Participants with at least one follow-up behavioral assessment visit were included in this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale | 2.6 (1.0) | 4.5 (1.6)

2. Primary Outcome: Change in Neuropsychiatric Inventory (NPI) Total Score Over the Course of Study Participation
Description: The Neuropsychiatric Inventory (NPI) is a 12-item scale that assesses the frequency and severity of behavioral symptoms in patients with dementia. Each Neuropsychiatric Inventory item ranges from 0 to 12. Therefore the Neuropsychiatric Inventory total score has a minimum total value of 0 and maximum 144, where 144 indicates higher levels of behavioral symptoms.
  A change in Neuropsychiatric Inventory total score that is a negative number (that is, an Neuropsychiatric Inventory score decrease), indicates behavioral improvement.
Time Frame: Weeks 2, 4, 6, and 8 (change from Baseline)
Population: Participants with at least one follow-up behavioral assessment visit were included in this analysis.
  The mean group change was calculated by calculating the mean of each participant's follow-up measures, subtracting this mean from the baseline value, and then from these values, calculating group means and standard deviations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale | -19 (21) | -2 (15)

3. Secondary Outcome: Number of Behavioral Assessment Visits Completed
Description: This measure reflects the length of time participants remained in the study. There were 6 behavioral assessment visits included in the protocol.
Time Frame: Last behavioral assessment (Baseline, Weeks 1, 2, 4, 6, or 8)
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 12 | 12
number of visits | 4.8 (1.6) | 4.5 (1.8)

4. Secondary Outcome: Change in Brief Psychiatric Rating Scale (BPRS) Total Score Over the Course of Study Participation
Description: The Brief Psychiatric Rating Scale (BPRS) is an 18-item scale that rates psychiatric symptoms. Each item ranges from 1 to 7. Therefore, the Brief Psychiatric Rating Scale total score ranges from a minimum of 0 to a maximum of 126, where 126 indicates higher levels of behavioral symptoms.
  A change Brief Psychiatric Rating Scale score that is a negative number (that is, a Brief Psychiatric Rating Scale score decrease), indicates behavioral improvement.
Time Frame: Weeks 2, 4, 6, and 8 (change from Baseline)
Population: Participants with at least one follow-up behavioral assessment visit were included in this analysis.
  The mean group change was determined by calculating the mean of each participant's follow-up measures, subtracting this mean from the baseline value, and then from these values, calculating group means and standard deviations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale | -9 (9) | -3 (5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from informed consent up until volunteers reached the end of their participation per protocol. Monitoring period was 10-12 weeks (2-4 weeks to start and titrate study drug, plus the 8 week follow-up period).
Description: Adverse effects were collected at each study visit. Study staff inquired about specific symptoms known to be potential side effects of prazosin using a preexisting checklist. Participants and their study companions were also asked about any new changes in health or medications.
Arm/Group | Prazosin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin (N=12) | Placebo (N=12)
sedation (Nervous system disorders) | 3 (3) | 3 (3)
confusion (Nervous system disorders) | 1 (1) | 4 (4)
lower extremity edema (Vascular disorders) | 1 (1) | 2 (2)
hypotension (Vascular disorders) | 2 (2) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
hallucinations (Psychiatric disorders) | 1 (1) | 1 (1)
dizziness on standing (Vascular disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No